CLINICAL TRIAL: NCT03258034
Title: Phase II Study of Convernsion Therapy Using S1/Paclitaxel Chemotherapy Plus Apatinib in ELM Gastric Cancer
Brief Title: A Feasibility Study for Convernsion Therapy Using S1/Paclitaxel Chemotherapy Plus Apatinib in ELM Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G328
Record Dates: First submitted 2017-08-20; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Gastric Cancer
Keywords: Conversion therapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conversion treatment (Experimental): after 3-4 cycles S1/Paclitaxel chemotherapy plus Apatinib,subsequent surgery will be conducted with curative intent.
  Interventions: Drug: SPA

INTERVENTIONS:
Drug: SPA — S1/Paclitaxel chemotherapy plus Apatinib S1:60mg twice daily(after the breakfast and supper) for two weeks, and then suspend for one week Paclitaxel:150mg/m2,iv, 3h, at day1 Apatinib:425mg once daily

SUMMARY:
The prognosis of Extensive lymph nodes metastatic(ELM) gastric cancer is poor. Chemotherapy occasionally converts it to a resectable cancer. Previous studies showed patients with ELM gastric cancer may obtain a survival benefit from chemotherapy and subsequent curative surgery. The key of conversion therapy of ELMGC is the high response rate. Apatinib, a novel targeted inhibitor of VEGF receptor 2 (VEGFR2), shows significant antitumor activity in the patients with GC. On the basis of our previous Ahead-G325 study, The purpose of this study is to investigate the efficacy and safety of S1/Paclitaxel chemotherapy plus Apatinib in the conversion therapys of ELM gastric cancer.

DETAILED DESCRIPTION:
The investigators will apply SPA regimen for coversional therapy to abtain high response rate. Paclitaxel：150 mg/m2 i.v.3h , given on the first day. Apatinib, oral ,initial dose :425mg, QD, after meal ( try to take the medicine at the same time of the day ). Dose adjustment: Down-regulate the dosage to 250 mg per day at the first time. If the patient totally recovers from the toxic reaction after the regulation, we could up-regulate the dosage back to the former level. If the downregulation occurs again according to the protocol , then the up-regulation will be forbidden.

S-1 dosage: According to the body surface area, the initial dosage of S-1 is decided by the following criteria. Take the medicine twice daily (after breakfast and supper) for 2 weeks, then suspend for 1 week. Preventive medication: To prevent serious allergic reaction of Paclitaxel, preventive medication should be given in advance. We usually give dexamethasone 20mg orally 12 and 6 hours before the Paclitaxel, and diphenhydramine (or something analogous) 50 mg, cimetidine 300mg (or ranitidine 50mg) I.V. 30-60 minutes before the Paclitaxel. Repeat the therapeutic schedule every 3 weeks. 3-4 cycles of neoadjuvant chemotherapy before surgery, stop Apatinib in the last cycle.4 cycles of adjuvant chemotherapy including S-1 and Apatinib 4 to 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ELM gastric cancer as proven histologically under following condition: unable radical excision due to the abdominal aorta a2-b1 or extensive lymph nodes metastatic,
* Definitely diagnosed as above stage of gastric cancer before operation via CT of MRI, ultrasonic endoscopy, PET-CT, or through the laparoscopic exploration if necessary
* Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy)
* Negative HER-2 state
* ECOG(Eastern Cooperative Oncology Group): 0~2
* Age: 18~70 years old- survival time > 3monts
* Normal hemodynamic indices before the recruitment(including blood cell count and liver/kidney function ). For example: WBC>4.0*109/ L, NE>1.5*109/L, PLT>100*109/L, BIL<1.5 times of upper limit of normal reference value, ALT and AST<2.5 times of upper limit of normal reference value, and CRE<1.2mg/dl
* Good cardiac function before the recruitment, no seizure of myocardial infarction in past half years, and controllable hypertension and other coronary heart disease
* Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver)
* Not participating in other clinical trials before and during the treatment
* Signed the Informed Consent Form
* No peritoneal metastatic and CY0 in 28 days by laparoscopic exploration
* Non-gastric stump cancer
* No esophagus infiltrating or infiltrating less than 3cm

Exclusion Criteria:

* Distal metastasis to Mediastinal lymph node,liver ,peritoneal,pleural effusion ,ascites,above 16a2-b1 and others
* Severe mental illness
* Her-2 positive, desire for hercptin treatment
* Ever administrated with other drugs(including TCM drugs) before the recruitment, or no guarantee of progress according to the study requirement after recruitment
* Allergy to the drugs in this protocol
* Pregnant and lactating women
* Women at childbearing age and of pregnancy desire during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-24 (Estimated); Primary Completion 2020-08-22 (Estimated); Study Completion 2021-10-22 (Estimated)

PRIMARY OUTCOMES:
3 year OS | 3 years
  The overall survival time

SECONDARY OUTCOMES:
radical resection rate | 4 months
  the radical resection rates
3 year DFS | 3 years
  the diesease free survival time
5 year OS | 5 years
  The overall survival time
adverse events | 7months
  number and degree of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, Study Director — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- The first affiliated hospital of zhejiang chinese medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No